CLINICAL TRIAL: NCT01513031
Title: Pilot Project to Determine Rates and Reasons for Non-Adherence in Patients Receiving Chronic Oral Antiarrhythmic Therapy for Atrial Fibrillation in the State of Nebraska
Brief Title: Determination of Rates and Reasons for Non-Adherence to Anti-Arrhythmic Therapy for Atrial Fibrillation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Creighton University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DRONE_L_06034; 11-16223 (Other: Institutional Review Board)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation; Medication Adherence
Keywords: Atrial fibrillation; Anti-arrhythmic medication; Medication adherence
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phone follow-up (Experimental): All study participants will be receiving education and monthly telephone follow-up.
  Interventions: Other: Education and telephone follow-up

INTERVENTIONS:
Other: Education and telephone follow-up — Education related to anti-arrhythmic therapy and monthly telephone follow-up to assess adherence to medication.

SUMMARY:
The purpose of this study is to determine if follow-up by a pharmacist over the telephone improves adherence and short term clinical outcomes in the patient with atrial fibrillation prescribed an oral anti-arrhythmic medication. This study will also identify the reasons people stop taking their anti-arrhythmic therapy. A pharmacist will provide medication counseling about their anti-arrhythmic therapy, then will follow-up by telephone on a monthly basis to assess adherence over one year.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed a new anti-arrhythmic medication for atrial fibrillation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adherence to anti-arrhythmic medication | 1 year
  Assessing whether patients stop taking anti-arrhythmic medication without instruction to do so by their physician.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Hilleman, PharmD, Principal Investigator — Creighton University
Locations (3):
- United States (3):
  - Bryan LGH, Lincoln, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska